CLINICAL TRIAL: NCT00129909
Title: Evaluation of a Primary Treatment Algorithm Using Fixed Dose Combination Therapy for the Management of Hypertension - Control and Intervention Arms
Brief Title: STITCH (Simplified Therapeutic Intervention To Control Hypertension)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Western Ontario, Canada (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RPO402A; RPO402B
Record Dates: First submitted 2005-08-10; First posted 2005-08-12 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Hypertension
Keywords: hypertension; family physicians; fixed dose combination therapy; cluster randomized controlled trial
MeSH Terms: conditions — Hypertension | interventions — Combined Modality Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: fixed dose combination therapy

SUMMARY:
The objective of this study is to assess whether the implementation of a primary treatment algorithm using a fixed dose combination therapy will improve the management of hypertension when compared to usual management.

DETAILED DESCRIPTION:
There is a clear need for improved approaches for both improved blood pressure control and improved compliance with medication regimens. Although decreasing the frequency of drug taking does improve blood pressure control, whether fixed-dose combinations are more effective than taking multiple tablets is unknown. Additionally, notwithstanding the presence of excellent evidence-based recommendations for the treatment of hypertension, the choices for practitioners in regards to first line therapy is widening (and may be more confusing, especially in the setting of the proliferation of recommendations for a range of diseases). Whether a simplified treatment algorithm, consistent with the Canadian Hypertension Education Program (CHEP) guidelines but using a step-care approach, might improve management of hypertension is unknown. The current study will determine the effectiveness of a simplified treatment algorithm which incorporates early use of a fixed-dose combination therapy.

This is a cluster randomized controlled trial. Approximately 50 family practices eligible for study participation will be randomized in a 1:1 ratio to implement a treatment algorithm or to continue usual care for the management of hypertension. The randomization schedule will be stratified by the year of graduation of the family physician (< 1984 or ≥ 1984). Within each practice, 50 subjects will be managed according to the algorithm or usual care and will be followed for six months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 years or older
* Hypertension SBP ≥ 140 mmHg or DBP ≥ 90 mmHg whether untreated or partially treated
* Absence of ischemic heart disease, atrial fibrillation, peripheral vascular disease, stroke and chronic kidney disease
* Not participating in other hypertension studies
* Ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2081 (Actual)
Dates: Start 2005-05; Primary Completion 2006-09 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
The primary measure of outcome is the proportion of subjects treated to target (systolic blood pressure [SBP] <140 mmHg and diastolic blood pressure [DBP] <90 mmHg) at 6 months, compared at the practice level.

SECONDARY OUTCOMES:
Secondary measures of response will include the change at 6 months in systolic blood pressure and diastolic blood pressure. These outcomes will be compared at the practice level
Provider satisfaction will be obtained by means of a questionnaire administered at each practice after the last study participant completes the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ross D Feldman, MD, Study Director — Western University, Canada
Locations (1):
- Robarts Research Institute, London, Ontario, Canada

REFERENCES:
- [Background] Kirkland SA, MacLean DR, Langille DB, Joffres MR, MacPherson KM, Andreou P. Knowledge and awareness of risk factors for cardiovascular disease among Canadians 55 to 74 years of age: results from the Canadian Heart Health Surveys, 1986-1992. CMAJ. 1999;161(8 Suppl):S10-6. PMID 10551207
- [Background] Berlowitz DR, Ash AS, Hickey EC, Friedman RH, Glickman M, Kader B, Moskowitz MA. Inadequate management of blood pressure in a hypertensive population. N Engl J Med. 1998 Dec 31;339(27):1957-63. doi: 10.1056/NEJM199812313392701. PMID 9869666
- [Background] Khan NA, McAlister FA, Campbell NR, Feldman RD, Rabkin S, Mahon J, Lewanczuk R, Zarnke KB, Hemmelgarn B, Lebel M, Levine M, Herbert C; Canadian Hypertension Education Program. The 2004 Canadian recommendations for the management of hypertension: Part II--Therapy. Can J Cardiol. 2004 Jan;20(1):41-54. PMID 14968142
- [Background] ALLHAT Officers and Coordinators for the ALLHAT Collaborative Research Group. The Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial. Major outcomes in high-risk hypertensive patients randomized to angiotensin-converting enzyme inhibitor or calcium channel blocker vs diuretic: The Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT). JAMA. 2002 Dec 18;288(23):2981-97. doi: 10.1001/jama.288.23.2981. PMID 12479763